**Document:** TDOC-0013927

Version: 5.0; Most-Recent; Effective; CURRENT  Status: Effective

## **Short Title:**

Effective Date: 05-Feb-2018

Biostatistics Safety Analysis Plan – C-09-043

## **Full Title:**

Biostatistics Safety Analysis Plan – C-09-043

Long Term Safety Protocol for AcrySof® CACHET® Phakic **Protocol Title:** 

Lens

25-5223/ NCT01497067 **Project Number:** 

**Reference Number:** PC2174.00

**Protocol TDOC Number:** TDOC-0010249

**Author:** 

See last page for electronic approvals. **Approvals:** 

**Job Notes:** 

C-09-043 is the extended safety follow-up study for subjects previously implanted with the AcrySof® CACHET® Phakic Lens (L-series) in clinical studies C-02-23, C-02-40, C-03-21 and C-05-57.

**Document:** TDOC-0013927

Version: 5.0; Most-Recent; Effective; CURRENT

 Status: Effective

Effective Date: 05-Feb-2018

# **Summary:**

# **Evaluability**

All subjects enrolled in the study will be considered evaluable for the safety analysis.

# **Analysis**

The primary objective is to estimate the annualized endothelial cell loss rate (for up to 10 years following date of implantation) of subjects previously implanted with the AcrySof® CACHET® Phakic Lens (L-Series) from clinical studies C-02-23, C-02-40, C-03-21 and C-05-57.

The secondary objective is to collect additional safety data that may identify risk factors for eyes with significant endothelial cell loss.

# **Safety Variables and Assessments**

The safety parameters include:

- Central Endothelial Cell Density
- Adverse Events



Version: 5.0; Most-Recent; Effective; CURRENT

Effective Date: 05-Feb-2018

Status: Effective 

# **Table of Contents**

| | 4 |
|--------------------------------------------------|----|
| | 4 |
| | 4 |
| | 4 |
| | 4 |
| 1. STUDY SUMMARY | 5 |
| 2. SAFETY VARIABLES | 7 |
| 2.1. Description | 7 |
| 2.2. Measurement Time. | 8 |
| 2.3. Unit of Analysis | 9 |
| 2.4. Descriptive Statistics | 9 |
| 3. DATA SETS ANALYZED | 9 |
| 3.1. Safety | 9 |
| 3.1.1. Evaluability Strategy | 9 |
| 3.1.2. Handling of Dropouts or Missing Data | 9 |
| 4. ANALYSIS OF SAFETY | 10 |
| 4.1. Maintenance of Endothelial Cell Density | 10 |
| 4.1.1. Description | 10 |
| 4.1.2. Endothelial Cell Loss over Time (Chronic) | 10 |
| | 11 |
| 4.2. Adverse Events | 15 |
| 4.2.1. Adverse Event Definitions | 15 |
| 4.2.2. Adverse Event Analysis | 15 |
| 5 Pafaranaas | 16 |

 Status: Effective

Effective Date: 05-Feb-2018

Status: Effective 

Effective Date: 05-Feb-2018

# 1. STUDY SUMMARY

| Study Phase: | | Not applicable – Study is observational only | |
|---|---|---|---|
| Test Article(s) / Product(s): | | AcrySof® CACHET® Phakic Lens (L-Series) | |
| Study Dosage / Us | | Intraocular lenses are implantable medical devices and are intended for long term use over the lifetime of the subject. The phakic intraocular lens may be removed as needed ( <i>e.g.</i> cataract extraction). | |
| Route of Administ | ration: | Not applicable | |
| Objective(s): | | The primary objective is to estimate the annualized endothelial cell loss rate (for up to 10 years following date of implantation) of subjects previously implanted with the AcrySof® CACHET® Phakic Lens (L-Series) from clinical studies C-02-23, C-02-40, C-03-21 and C-05-57. The secondary objective is to collect additional safety data that may identify risk factors for eyes with significant endothelial cell loss. | |
| Study Population: | | Subjects previously implanted with the AcrySof® CACHET® Phakic Lens (L-series) in clinical studies C-02-23, C-02-40, C-03-21 and C-05-57 (includes subjects who have had the lens explanted for any reason). | |
| Structure: | Parallel C | Group | Duration of Treatment: |
| | | | Duration of Assessment: |
| | Crossove | r | Number of Treatments: Number of Sequences: |
| | | | Number of Periods: |
| | | | Duration of Periods: |
| | | | Washout Between Yes No Periods: |
| | X Other | | No control, open label study |
| | | | Duration of Treatment: Subjects to be followed for 5 to 7 years (10 years from the time of implantation). |
| Multi-center: | X Yes No | Num | aber of Centers: Up to 35 |

Version: 5.0; Most-Recent; Effective; CURRENT **Document:** TDOC-0013927

 Status: Effective Masking: None Observer-Masked Patient-Masked Double-Masked Randomization: Group Assignment Ratio: Yes X No Concurrent None Control: No Treatment Placebo Active Specify: Specify: Other Estimated Total Sample Size: Required: N/A Planned: Up to 1321 eyes Safety **Primary Safety** Central endothelial cell density Variable(s): Adverse Events Adverse Events: Both volunteered and elicited

Effective Date: 05-Feb-2018

Print Date: Printed By:

Other:

**Document:** TDOC-0013927

Version: 5.0; Most-Recent; Effective; CURRENT  Status: Effective

Effective Date: 05-Feb-2018

# 2. SAFETY VARIABLES

# 2.1. Description

The safety of the AcrySof® CACHET® Phakic Lens (L-Series) will be assessed for the following safety parameters:

- Central Endothelial Cell Density
- Adverse Events



Table 2.2.-1: Study Plan


| Document: T | | -0013927 | Version | : 5.0 | ; Most-Recent; Effective; CURRI | ENT |
|---|---|---|---|---|---|---|
| Status: Effect | ıve | Year<br>10/10A | Day 3619 – 3740 | X | | X |
| | | Year<br>9.5/9.5A | Day 3436 – 3557 | X | | X |
| | | Year<br>9/9A | Day 3254 – 3375 | X | | X |
| | Nominal Time ± Visit Window Limits | Year<br>8.5/8.5A | Day 3071 – 3192 | X | | X |
| | | Year<br>8/8A | Day 2889 – 3010 | X | | X |
| | | Year<br>7.5/7.5A | Day 2706 – 2827 | X | | X |
| g | | Year<br>7/7A | Day 2524 – 2645 | X | | X |
| Table 2.21: Study Plan | | Year<br>6.5/6.5A | Day 2341 – 2462 | X | | X |
| 2.21: | | Year<br>6/6A | Day 2159 – 2280 | X | | X |
| Table | | Year<br>5.5/5.5A | Day 1976 – 2097 | X | | X |
| | | Year<br>5/5A | Day 1794 – 1915 | X | | X |
| | | Year<br>4/4A° | Day <sup>b</sup> 1429 – 1550 | X | | X |
| | | Entrance<br>Visit <sup>a</sup> | | | | |
| ime | | | ent | ECD | | |
| .2. Measurement Time | | | Procedure / Assessment | | | Adverse Events |
| .2. Meas | | | Procedu | Central | | Adverse |

The subject's initial C-09-043 study examination may be Form 9 or later (i.e., Form 9, 10, 11, etc.). Point of entry is determined by each subject's eye surgery date and the next available visit listed here to enable continued yearly examination. As in previous studies, subjects with the AcrySof® CACHET® Phakic Lens (L-Series) implanted in both eyes will have separate study visits, as needed, for each eye to capture the data within the window of the annual implant date anniversary.

Study Day is relative to the surgery date for each implanted eye. þ

Data from subject's 2nd implant surgery will be captured on Forms designated with an "A".

**Document:** TDOC-0013927

Status: Effective 

Version: 5.0; Most-Recent; Effective; CURRENT

Effective Date: 05-Feb-2018

## 2.3. Unit of Analysis

The eye will be the unit of analysis for all safety parameters except for non-ocular adverse events where the unit of analysis will be subject.

## 2.4. Descriptive Statistics

Descriptive statistics for both eyes combined will be provided for endothelial cell density and adverse events. The statistics presented for continuous variables will include mean, median, standard deviation, number of eyes, minimum and maximum. The statistics for categorical variables will include sample size and percentage in the categories.

#### 3. DATA SETS ANALYZED

## 3.1. Safety

#### 3.1.1. EVALUABILITY STRATEGY

All subjects enrolled in the study will be considered evaluable for the safety analysis. All data collected in the study will be considered evaluable for the safety analysis with one exception. For subjects who have their AcrySof® CACHET® L-series Phakic Lens explanted and not replaced with another AcrySof® CACHET® L-series Phakic Lens, the post-explantation endothelial cell density data will be excluded from the statistical analyses other than a post-explant endothelial cell loss analysis. The post-explantation data will be used in subject narratives. The final evaluability (exclusion of post-explantation endothelial cell density data) will be determined prior to database lock.

## 3.1.2. HANDLING OF DROPOUTS OR MISSING DATA

All data will be used in the analyses. No imputation will be carried out for missing data.

Status: Effective 

Effective Date: 05-Feb-2018

#### 4. ANALYSIS OF SAFETY

# 4.1. Maintenance of Endothelial Cell Density

#### 4.1.1. DESCRIPTION

Endothelial cell density will be collected centrally . Three images at the center of the cornea are planned. Data reported on the CRF by the central reading center will include endothelial cell density and number of cells that were analyzed for each analyzable image. All recorded data from images will be used in the analysis. Although the central reading center will record the data separately for each image, the average cell density of the analyzable images for an individual eye for each corneal location (central ) will be used in all summary analyses.

# 4.1.2. ENDOTHELIAL CELL LOSS OVER TIME (CHRONIC)

Chronic endothelial cell loss is defined as loss from the Day 147-182 (Form 5 or 5A) visit (in the previous studies) to any subsequent visit.

## 4.1.2.1. CHRONIC CHANGE FROM DAY 147-182 (MONTH 6 IN PREVIOUS STUDIES)

Descriptive statistics will be provided for each scheduled visit, for endothelial cell density, for all eyes combined. The statistics presented for endothelial cell density (using the average from the analyzable images for each eye) will include mean, median, standard deviation, sample size, minimum, and maximum.

The percent change of mean endothelial cell density over time from Day 147-182 (Form 5 or 5A) in the previous studies to each visit in the current study will be calculated. The actual and annualized percent change of mean endothelial cell density from the Day 147-182 (Form 5 or 5A) exam to each scheduled visit in this study will be calculated and presented along with median, standard deviation, sample size, minimum and maximum. Tables presenting the mean, median, standard deviation, sample size, minimum and maximum of baseline (Form 5 or 5A in previous studies) endothelial cell density and cell density change from baseline to each scheduled visit in this study will be presented for all eyes combined.

Status: Effective 

Effective Date: 05-Feb-2018

## 4.1.2.2. POSTOPERATIVE CHANGE FROM PREOPERATIVE BASELINE

Descriptive statistics will be provided for change from preoperative baseline (in previous studies) to each scheduled visit in this study, for central endothelial cell density, for all eyes combined. The statistics presented will include mean, median, standard deviation, sample size, minimum and maximum. The percent change of mean endothelial cell density from preoperative baseline (Form 0 or 0A in previous study) to each scheduled postoperative visit (both in previous studies and this study) will be calculated to determine subjects who had  $\geq 30\%$  loss. A table showing the number and percent of eyes which had the onset of  $\geq 30\%$  endothelial cell loss (central of  $\leq 1500$  endothelial cells/mm² (occurring 6 months or later following implantation) will be presented.

In addition, the mean actual and annualized percent change of endothelial cell density (using the average from the analyzable images for each eye) of all subjects from baseline to each visit will be calculated and presented along with median, standard deviation, sample size, minimum and maximum. These tables will be presented for all eyes combined.



**Document:** TDOC-0013927

Version: 5.0; Most-Recent; Effective; CURRENT

Effective Date: 05-Feb-2018

Status: Effective 

Status: Effective 

Effective Date: 05-Feb-2018

Status: Effective 

Effective Date: 05-Feb-2018

Status: Effective 

Effective Date: 05-Feb-2018



# 4.2. Adverse Events

## 4.2.1. ADVERSE EVENT DEFINITIONS

Adverse events (AE), serious adverse events (SAE), adverse device effects (ADE), are defined as set forth in Section 12.1. of the protocol.

## 4.2.2. ADVERSE EVENT ANALYSIS

Adverse events will be coded with MedDRA Preferred Term codes. Descriptive statistics (number and percent of eyes) will be presented for each MedDRA Preferred Term category of ocular adverse events and serious ocular adverse events reported, separately for first

**Document:** TDOC-0013927 **Version:** 5.0; Most-Recent; Effective; CURRENT

Status: Effective 

Effective Date: 05-Feb-2018

implanted eye, second implanted eye and both eyes combined. Separate tables will be generated for AEs, SAEs, and ADEs. Descriptive statistics (number and percent of subjects) will be presented for each MedDRA Preferred Term category and System Organ Class of non-ocular adverse events and serious non-ocular adverse events reported. In addition, a one-sided upper 95% confidence interval on the percent of each MedDRA Preferred Term code will be calculated



A listing of all adverse events and serious adverse events including investigator, subject number, onset day, eye, lens model, causality assessment, severity, outcome and the MedDRA Preferred Term code for the adverse event will also be provided.

### 5. References

<sup>1</sup>Zarr, JH. Biostatistical Analysis. 3rd ed. Upper Saddle River, New Jersey: Prentice-Hall, Inc;1996: 525-526.

<sup>2</sup>SAS Help and Documentation (SAS Version 9.4). The FREQ Procedure-Binomial Proportion-Wald Confidence Limits.

**Document:** TDOC-0013927

Version: 5.0; Most-Recent; Effective; CURRENT

Effective Date: 05-Feb-2018

Status: Effective

| Date/Time | Ciana ad have | Lucatific antique |
|---------------------|---------------|-------------------|
| (mm/dd/yyyy GMT): | Signed by: | Justification: |
| 01/30/2018 21:15:21 | t | Statistician |
| 01/30/2018 21:57:06 | | Biostatistics |
| 01/31/2018 15:47:28 | | Medical Safety |
| 02/02/2018 21:59:43 | | Clinical Lead |